CLINICAL TRIAL: NCT03991182
Title: Evaluation of Scaling Up Early Childhood Development in Zambia
Acronym: SUpErCDZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Right to Care Zambia (RTCZ) (Unknown); Swiss Tropical & Public Health Institute (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Grand Challenges Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38950; TTS-1802-21377 (Other Grant/Funding Number: Grand Challenges Canada); 72061119FA00001 (Other Grant/Funding Number: United States Agency for International Development (USAID))
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Early Childhood Development
Keywords: Community based parenting; Developmental outcomes; Maternity waiting homes (MWHs); Safe Motherhood Action Group leaders (SMAGs); Zambia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-based parenting group (Experimental): The community-based parenting group will include 39 health zones and 585 caregiver-child dyads
  Interventions: Other: SMAGs trained on ECD curriculum; Other: Head women trained on ECD curriculum; Behavioral: Head women led parent groups
- Control group (Active Comparator): The control group will include 39 health zones and 585 caregiver-child dyads
  Interventions: Other: Usual care of children 0-5 months

INTERVENTIONS:
Other: SMAGs trained on ECD curriculum — 50 volunteers (primarily SMAGs- Safe Motherhood Action Group members) associated with the health facility will be trained using a training -of-trainers approach on the e ECD (early childhood development) curriculum
  Arms: Community-based parenting group
Other: Head women trained on ECD curriculum — Each of the 50 trained SMAGs will train 10 head women on the ECD curriculum
  Arms: Community-based parenting group
Behavioral: Head women led parent groups — Every two weeks 500 trained head women lead parent group meetings on childhood development and nutrition to caregiver-child dyads
  Arms: Community-based parenting group
Other: Usual care of children 0-5 months — The traditional care and education of caregivers/parents for children 0-5 months
  Arms: Control group

SUMMARY:
In Zambia, 40% of children under five years of age are stunted and 6% are wasted. While the Zambian government has focused on child nutrition in recent years, more focus on holistically improving early child development (ECD) is needed. Through a previous randomized controlled trial, the investigators developed a community-based parenting intervention and demonstrated that this intervention can improve children's developmental outcomes in Zambia, including nutritional status and their early language development. During fortnightly group meetings, parents learn a diverse curriculum that includes content on: 1) cognitive stimulation and play practices; 2) child nutrition and cooking practices; and 3) self-care for good mental health. This information and learning content is delivered by supervised community volunteers using an interactive theatre-based approach.

In this study, the newly established maternity waiting homes (MWHs) and affiliated Safe Motherhood Action Group leaders (SMAGs) will be used as a novel platform to launch and support community-based parenting groups, embedding this program directly into the existing health system, and making them more feasible for scale-up and sustainability.

Despite the positive impact of the proposed parenting-group model in the pilot trial, this model is not currently operating in Zambia. By integrating this intervention into the existing health system, large populations of rural children exposed to high levels of adversity in the critical early years of life could be reached in a nationally scalable fashion. As part of this project, the investigators propose to implement and rigorously assess the impact of this approach in four districts of Zambia.

DETAILED DESCRIPTION:
This research will utilize a cluster-randomized controlled trial with integrated mixed-methods process evaluation to understand the impact of parenting groups on child development outcomes when delivered at scale. The specific objectives are to: 1) assess the impact of the intervention on early childhood development outcomes; 2) assess the degree to which the intervention was implemented according to the project plan and to document adjustments made during the course of the project; 3) describe and document the perceptions of caregivers on parent groups, as well as any behavioral changes in parenting or in mother support networks resulting from participating in parenting groups; and approaches to achieving caregiving gender equality at household level; and, 4) generate a set of recommendations for the Government of the Republic of Zambia to further adapt and/or scale up community parenting groups based on the summative findings from this study.

For the impact evaluation the investigators will collect data from two main sources: 1) Household Surveys and 2) In-depth interviews at both baseline and endline data collection. In addition, at endline we will assess child development using the Malawi Developmental Assessment Tool (MDAT).

For the process evaluation, the investigators will conduct record review of parenting groups attendance registers and SMAG log books. The investigators will conduct in-depth interviews with health systems staff (province, district and health facility), SMAGs, and head women from all intervention sites, and focus group discussions with caregivers who meet the study eligibility criteria in both intervention and control zones.

ELIGIBILITY:
Caregiver-child dyads in the impact cohort

Inclusion Criteria:

* Children aged 0-5 months at baseline in the catchment areas of the ten selected health facilities in Southern and Eastern Provinces will be eligible to participate
* Child's primary caregiver must be 15 years or older
* Child's primary caregiver must be a female (because the participants in the women's group may feel uncomfortable discussing certain issues if a man is present)

Exclusion Criteria:

* Caregivers who are unwilling to provide informed consent
* Families that plan to move from their health center catchment zone during the period of the study

In-depth interviews (IDI)

Inclusion Criteria:

* A member of the health facility staff at a study site for at least 6 months; or
* A district or provincial level health staff; or
* A SMAG member at a study site who has been trained to implement the parenting group intervention; or
* A 'head mother' leading parenting group sessions within their communities; and ≥18 years of age and provided informed consent to participate in the IDI.

Exclusion criteria

-None

Focus group discussions (FGDs)

Inclusion Criteria:

* A woman or a man with child under 3 years of age; or
* Community health volunteers [SMAG, community health worker (CHW) or TBA]; and
* Resident within the project zones; and -≥18 years of age

Exclusion Criteria:

-None

Min Age: 0 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1108 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Child linear growth: Stunting | Children aged 0-5 months at baseline (August-September 2019) and end line (September 2021), child aged 24-29 months
  Heights of all study children will be measured. Height-for-age z-scores will be calculated using standard World Health Organization (WHO) criteria. Stunting will be defined as having a height-for-age z-score < -2. The difference in the prevalence of stunting between children in the intervention and comparison areas will be determined.
Child development z-scores based on Malawi Developmental Assessment Tool (MDAT) | At endline (child aged 24-29 months) children are assessed using the MDAT. Scores are standardized within the study sample for analysis.
  Cognitive function measurements
Caregiver Reported Early Development Index | Children aged 0-5 months at baseline (August-September 2019) and end line (September 2021), child aged 24-29 months
  Summary score of child development measures (motor, cognitive, language, and social emotional skills)

SECONDARY OUTCOMES:
Proportion of children receiving all age-appropriate vaccines | Baseline (child 0-5 months), Endline (child aged 24-29 months)
  We will collect data at baseline and endline on whether the study children are up to date on vaccines as recommended by the government vaccination schedule.
Proportion of children receiving vitamin A supplementation | Baseline (child 0-5 months), Endline (child aged 24-29 months)
  Caregivers will be asked about vitamin A supplementation and responses will be compared to child development outcomes
Number of well-baby visits attended | Baseline (child 0-5 months), Endline (child aged 24-29 months)
  Caregivers will be asked about the health seeking behaviors for the child; results will be compared against government recommendations and against child development outcomes
Average time spent reading with the child | Baseline (child 0-5 months), Endline (child aged 24-29 months)
  Caregivers will be asked about their engagement with the child and other adult engagement with the child at baseline and endline
Average time spent playing with the child | Baseline (child 0-5 months), Endline (child aged 24-29 months)
  Caregivers will be asked about their engagement with the child and other adult engagement with the child at baseline and endline

OTHER OUTCOMES:
Child diet diversity | Baseline (child 0-5 months), Endline (child aged 24-29 months)
  Caregivers will be asked about child feeding habits and dietary diversity
Caregiver mental health based on the Self Reporting Questionnaire 20-item (SRQ-20) | Baseline (child 0-5 months), Endline (child aged 24-29 months)
  Caregivers will be asked a series of questions on their personal mental health using an instrument that has been adapted to the context

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Scott, DrPH MPH, Principal Investigator — Boston University; Thandiwe Ngoma, Principal Investigator — Right to Care - Zambia
Locations (3):
- Zambia (3):
  - Nyimba District Medical Office, Nyimba, Eastern Province
  - Choma District Medical Office, Choma, Southern Province
  - Kalomo District Medical Office, Kalomo, Southern Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rockers PC, Zanolini A, Banda B, Chipili MM, Hughes RC, Hamer DH, Fink G. Two-year impact of community-based health screening and parenting groups on child development in Zambia: Follow-up to a cluster-randomized controlled trial. PLoS Med. 2018 Apr 24;15(4):e1002555. doi: 10.1371/journal.pmed.1002555. eCollection 2018 Apr. PMID 29689045
- [Background] Rockers PC, Fink G, Zanolini A, Banda B, Biemba G, Sullivan C, Mutembo S, Silavwe V, Hamer DH. Impact of a community-based package of interventions on child development in Zambia: a cluster-randomised controlled trial. BMJ Glob Health. 2016 Nov 22;1(3):e000104. doi: 10.1136/bmjgh-2016-000104. eCollection 2016. PMID 28588962
- [Background] Scott NA, Kaiser JL, Vian T, Bonawitz R, Fong RM, Ngoma T, Biemba G, Boyd CJ, Lori JR, Hamer DH, Rockers PC. Impact of maternity waiting homes on facility delivery among remote households in Zambia: protocol for a quasiexperimental, mixed-methods study. BMJ Open. 2018 Aug 10;8(8):e022224. doi: 10.1136/bmjopen-2018-022224. PMID 30099401

DOCUMENTS (1):
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT03991182/ICF_000.pdf